CLINICAL TRIAL: NCT02811848
Title: Pilot Feasibility Study: Recruiting African American Fathers and Their Adolescent Sons for Qualitative, Sexual Health Research
Brief Title: Recruiting African American Fathers/ Sons
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00071686
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Sexually Transmitted Diseases; HIV
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barbers: Barbers that service African American clientele mainly will be recruited for this study; there is no intervention.

SUMMARY:
The purpose of this study is to develop and pilot test recruitment methods for a future study of prevention of sexually transmitted infections (STI), including the human immunodeficiency virus (HIV), among Black adolescent boys through sexual health education by their fathers.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs), including the human immunodeficiency virus (HIV), are a health problem for all adolescents, regardless of race. Presently, there are nearly 110 million cases of sexually transmitted infections (STI) in the United States. Annually, there are more than 19.7 million new STI cases, of which half are accounted for by youth. Of those, more than half are accounted for by youth ages 15 to 24 years. However, Black males between the ages of 13 and 17 are disproportionately affected by STIs such as chlamydia, gonorrhea, syphilis, and HIV/AIDS; they currently account for 50% of HIV infections among all youth. Additionally, the rate of HIV infection among young black gay or bisexual men is twice that of young white men. Researchers have pointed to the need to involve Black men who are fathers in interventions to decrease the epidemic of STIs and HIV among Black adolescent boys. However, youth-focused interventions from the Centers for Disease Control and Prevention (CDC) include only one intervention with a focus on the father and son as a dyad. Thus more research is clearly needed with this focus, but challenges with recruitment need to first be addressed. Challenges in recruiting Black men for health research are reflected in efforts by the National Institutes of Health (NIH) to promote research that includes minorities and in particular Black fathers. Barriers to research participation include ongoing distrust of health researchers because of the historic failing of the medical field in the Tuskegee syphilis study of rural Black men; this occurred more than 47 years ago but still remains important today. Barriers also include lack of knowledge of the benefits of research. Because of this lack of participation of Black men in research we have only limited understanding of their perceptions of many health issues. In order to involve this population in research, barriers and challenges to their involvement must be overcome. One way to begin this is to engage with leaders in their communities, to effectively communicate research objectives and begin building trusting relationships. Establishing relationships with community leaders can facilitate recruitment in research and help to overcome some of the barriers and challenges for Black men. Important elements of building those relationships include discussing research procedures, hypotheses, pilot data, and plans to bring results of research back to the community for future utilization. This proposed study will therefore seek to implement these elements of trust with local barbers and barbershops. In the Black community, barbers have been identified as community leaders and a great recruiting source for work on health promotion and disease prevention in the areas of hypertension and prostate cancer. However, few studies have used barbershops for sexual health related content focusing on Black fathers and their adolescent boys.

To create a successful recruitment process for Black men and their sons, a strategic plan of action is necessary prior to implementing a study. The first step is to gain a deeper understanding of effective strategies to include Black men in research. Therefore, the proposed pilot study will develop and test the feasibility of a recruitment process for Black men who are fathers and their adolescent sons, using barbershops and barbers as recruiters and advocates. Barbers will be assessed for their willingness to serve as recruiters and advocates for sexual health related studies involving Black fathers and their adolescent sons, and their ideas for recruitment for this group. With this information we will develop and pilot a recruitment strategy, to be used in a future qualitative study: Assessing Black fathers' attitudes towards discussing sexual health with their adolescent son and Assessing Black adolescent boys' attitudes towards their father as a sexual health educator. This future study will identify fathers' attitudes towards their adolescent sons and sex and major influences on sexual behaviors of adolescent boys, identify fathers' perspectives on what and who is important to include in an intervention focused on STI and HIV prevention, develop a survey tool to assess a larger sample of African American fathers for a future study, and gain adolescent males' perspectives on the role of their fathers in their sexual health. Research has suggested that clear communication between Black parents and their youth about sexual health is associated with higher rates of sexual abstinence, condom use, and intent to delay initiation of sexual intercourse, which can prevent infectious diseases. However, barriers exist for parents in educating their youth about sexual health, including lack of knowledge and discomfort in talking about safe sex. Further, little research has been conducted specifically on the parental role of Black fathers in educating their sons. This study will identify the best strategies for recruiting Black fathers and their sons for research on the parental role of Black fathers in helping their sons avoid risky sex.

ELIGIBILITY:
* barbershop inclusion includes:

  * serving a predominantly young to middle age, Black clientele
  * willingness to recruit barbers at each shop to participate in a 2-hour focus group session.
* Inclusion criteria for barbers:

  * a full time barber
  * age 18 years or older
  * willing to participate in a 2-hour focus group session
  * able to provide written consent
  * serving primarily young to middle age Black males.
* Fathers are selected by the following inclusion criteria:

  * self-identification as Black or African American
  * father of an adolescent male child age 11-18 (father in this study will be defined as biological father, stepfather, or father by adoption)
  * residence in or outside of the home
  * a consistent relationship with son (defined as communicating with son at least weekly)
  * willingness to participate in a 2-hour focus group session, and written consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Barbers who serve majority African American fathers and male youth.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Recruitment Strategy for the recruitment of African American father/son dyads | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Schenita Randolph, Principal Investigator — Duke University School of Nursing
Locations (1):
- Barbershops, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided